CLINICAL TRIAL: NCT05683548
Title: Compassionate Use Access to REP 2139-Mg for the Treatment of Chronic HBV Infection or Chronic HBV / HDV Co-infection
Brief Title: Replicor Compassionate Access Program
Acronym: RCAP
Status: No longer available | Type: Expanded Access
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RCAP
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Viral Hepatitis B; Viral Hepatitis D; Cirrhosis, Liver; Decompensated Cirrhosis; Ascites Hepatic; Varices, Esophageal; Hepatocellular Carcinoma
Keywords: nucleic acid polymer; REP 2139-Mg; HBV; HDV; cirrhosis; functional cure
MeSH Terms: conditions — Hepatitis B; Hepatitis D; Liver Cirrhosis; Esophageal and Gastric Varices; Carcinoma, Hepatocellular; Fibrosis | interventions — Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: REP 2139-Mg — REP 2139-Mg is the magnesium chelate complex of REP 2139
Drug: Tenofovir Disoproxil Fumarate
  Other Names: Viread
Drug: Pegylated interferon alpha2a
  Other Names: Pegasys

SUMMARY:
The goal of this compassionate access program is to provide early access to REP 2139-Mg for patients with HBV mono-infection or HBV / HDV co-infection who either have advanced (decompensated) cirrhosis or who have failed to response to other other antiviral agents either approved or under development and who are in danger of progressing to decompensated cirrhosis.

This compassionate access program will provide access to a once weekly regimen of subcutaneously (SC) administered REP 2139-Mg for a period of 48 weeks with the goal of achieving functional cure of HDV and or HBV, with the reversal of liver disease in the absence of antiviral therapy. The safety, tolerability and efficacy of SC REP 2139-Mg will be monitored during and after therapy

DETAILED DESCRIPTION:
Nucleic acid polymers (NAPs) block the assembly of hepatitis B virus (HBV) subviral particles and bind to the small and large hepatitis delta virus (HDV) antigen. In chronic HBV mono-infection, this leads to rapid HBsAg loss and in chronic HBV / HDV co-infection, simultaneous loss of HBsAg and HDV RNA. NAP-based combination therapy (using REP 2139-Mg) achieves high rates of functional cure of HBV and HDV in the absence of therapy in previous clinical trials limited to patients without cirrhosis.

The Replicor compassionate access program (RCAP) provides early access to individuals which have HBV mono-infection, or HBV / HDV co-infection who have not responded to existing approved or experimental therapies and are in danger of progressing advanced liver disease or who have already progressed to decompensated cirrhosis. Examples of previous therapy includes but is not limited to pegylated interferon (pegIFN), bulevirtide or lonafarnib.

Participants with failure to previous therapy with compensated cirrhosis will receive REP 2139-Mg (250mg SC qW), TDF (300mg PO QD) and pegIFN (90ug SC qW) for 48 weeks. Participants with decompensated cirrhosis will receive REP 2139-Mg (250mg SC qW) and TDF (300mg PO QD).

During therapy, safety will be monitored weekly and efficacy every 4 weeks.

Patients who maintain HBsAg loss for 6 months following removal of REP 2139-Mg and pegIFN will be eligible for removal of the remaining TDF therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HBV or HBV / HDV co-infection.
2. Prior failure to pegIFN, bulevirtide, or lonafarnib or combinations thereof with advanced fibrosis or compensated cirrhosis.
3. Decompensated cirrhosis.
4. Willingness to utilize adequate contraception while being treated with REP 2139-Mg and for 6 months following the end of REP 2139-Mg treatment.

Exclusion Criteria:

1. Women with positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG).
2. Breast-feeding women.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (13):
- Medical University of Vienna, Vienna, Austria
- France (9):
  - AP-HP Hôpital Beaujon, Clichy
  - CHU Lille, Lille
  - CHU-Limoges, Limoges
  - Hôpital Saint-Joseph, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CHU de Montpellier, Montpellier
  - Centre Hospitalier de Perpignan, Perpignan
  - CHU de Rennes, Rennes
  - CHU Rangueil, Université Toulouse 3, Toulouse
- Soroka Medical Center, Beersheba, Israel
- Padua University Hospital, Padua, Italy
- Koç University Medical School, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Vaillant A. REP 2139: Antiviral Mechanisms and Applications in Achieving Functional Control of HBV and HDV Infection. ACS Infect Dis. 2019 May 10;5(5):675-687. doi: 10.1021/acsinfecdis.8b00156. Epub 2018 Oct 5. PMID 30199230
- [Background] Blanchet M, Sinnathamby V, Vaillant A, Labonte P. Inhibition of HBsAg secretion by nucleic acid polymers in HepG2.2.15 cells. Antiviral Res. 2019 Apr;164:97-105. doi: 10.1016/j.antiviral.2019.02.009. Epub 2019 Feb 13. PMID 30771404
- [Background] Boulon R, Blanchet M, Lemasson M, Vaillant A, Labonte P. Characterization of the antiviral effects of REP 2139 on the HBV lifecycle in vitro. Antiviral Res. 2020 Nov;183:104853. doi: 10.1016/j.antiviral.2020.104853. Epub 2020 Jun 23. PMID 32585322
- [Background] Bazinet M, Pantea V, Cebotarescu V, Cojuhari L, Jimbei P, Albrecht J, Schmid P, Le Gal F, Gordien E, Krawczyk A, Mijocevic H, Karimzadeh H, Roggendorf M, Vaillant A. Safety and efficacy of REP 2139 and pegylated interferon alfa-2a for treatment-naive patients with chronic hepatitis B virus and hepatitis D virus co-infection (REP 301 and REP 301-LTF): a non-randomised, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2017 Dec;2(12):877-889. doi: 10.1016/S2468-1253(17)30288-1. Epub 2017 Sep 28. PMID 28964701
- [Background] Bazinet M, Pantea V, Cebotarescu V, Cojuhari L, Jimbei P, Anderson M, Gersch J, Holzmayer V, Elsner C, Krawczyk A, Kuhns MC, Cloherty G, Dittmer U, Vaillant A. Persistent Control of Hepatitis B Virus and Hepatitis Delta Virus Infection Following REP 2139-Ca and Pegylated Interferon Therapy in Chronic Hepatitis B Virus/Hepatitis Delta Virus Coinfection. Hepatol Commun. 2020 Nov 13;5(2):189-202. doi: 10.1002/hep4.1633. eCollection 2021 Feb. PMID 33553968
- [Background] Bazinet M, Pantea V, Placinta G, Moscalu I, Cebotarescu V, Cojuhari L, Jimbei P, Iarovoi L, Smesnoi V, Musteata T, Jucov A, Dittmer U, Krawczyk A, Vaillant A. Safety and Efficacy of 48 Weeks REP 2139 or REP 2165, Tenofovir Disoproxil, and Pegylated Interferon Alfa-2a in Patients With Chronic HBV Infection Naive to Nucleos(t)ide Therapy. Gastroenterology. 2020 Jun;158(8):2180-2194. doi: 10.1053/j.gastro.2020.02.058. Epub 2020 Mar 6. PMID 32147484
- [Derived] Stern C, Loustaud-Ratti V, Yurdaydin C, Brancaccio G, Jachs M, Reiberger T, Bardou-Jacquet E, Metivier S, Alric L, Colombain L, Meszaros M, Mathurin P, Yardeni D, Etzion O, Neumann-Haefelin C, Douglas M, Poulin S, Bazinet M, Metin RO, Vitale A, Gaeta GB, Schwarz M, Ben-Ali S, Bedoya JU, Testoni B, Zoulim F, Plissonnier ML, Levrero M, Paradis V, Francois S, de Freitas C, Kaysin F, Lecomte L, Morvan C, Schramko J, Bondezi K, Baril ME, Brichler S, Gerber A, Gordien E, Mackiewicz V, Dahari H, Svicher V, Chevaliez S, Vaillant A, Bourliere M. Safety and efficacy of REP 2139-Mg in patients with HDV-related advanced liver disease in an international compassionate access program. J Hepatol. 2025 Nov 6:S0168-8278(25)02612-1. doi: 10.1016/j.jhep.2025.10.029. Online ahead of print. PMID 41205755
- See also: Repicor Inc. — http://www.replicor.com
- See also: Interaction of NAPs with HDAg — http://www.replicor.com/wp-content/uploads/2020/12/NAPs-HDAg-interaction-AASLD-2017-poster-942.pdf